CLINICAL TRIAL: NCT02661386
Title: Esophageal Manometry During Recovery From Anesthesia: Pilot Study
Acronym: EMAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-15466
Record Dates: First submitted 2016-01-19; First posted 2016-01-22 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Motility Function

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Manometry Device (Other): During the last 10 minutes of subjects "waking up" from anesthesia, the motility procedure will be performed.
  Interventions: Device: Motility Procedure

INTERVENTIONS:
Device: Motility Procedure — The use of esophageal manometry device during general anesthesia

SUMMARY:
1. An intact pharyngoesophageal reflex is essential to protect the upper airway from aspiration of either mouth contents or regurgitated gastric refluxate. This reflex is essential at protecting the airway in all patients.
2. In patients, while under general anesthesia, it is postulated that an identifiable upper esophageal sphincter and esophageal peristalsis are not present.
3. With the cessation of general anesthetics, accompanied by the reversal of nerve block, normal pharyngoesophageal peristaltic activity correlates with awakening the patient from anesthesia. This would be identified by the performance of esophageal manometry.
4. A return of normal verbally stimulated pharyngoesophageal swallowing sequence accurately identifies a safe time to remove endotracheal tubes and/or reverse anesthesia. This verbally stimulated swallowing sequence correlated precisely with the return of objective pharyngoesophageal function.

DETAILED DESCRIPTION:
This pilot study will examine esophageal manometry in patients emerging from routine general anesthesia. Manometry of the esophagus is not a standard part of surgery or general anesthesia. The investigators will be using standard solid state high resolution manometry. One of the authors (JPC) evaluates all routine manometry for patients undergoing such procedures at both UCSF and SFGH. The use of manometry in patients recovering from anesthesia will permit the investigators to assess the recovery of a normal swallowing mechanism. An adequate determination of return of normal swallowing sequence is likely to determine the safe time for extubation. The investigators propose to, as a research study, investigate esophageal motor function using standard high resolution esophageal manometry in 10 patients recovering from general anesthesia. These studies are likely to document that the return of normal pharyngoesophageal function will coordinate with verbal commands to initiate swallowing. This pilot study will help clarify the precise timing of the return of normal function in the oropharynx and the proximal esophagus and thus determine the safe time for removal of the endotracheal or nasotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age (ASA I or II).
* Already scheduled for routine general anesthetic procedure requiring an endotracheal tube for anesthesia administration.
* Scheduled abdominal surgical procedure including endoscopy, colonoscopy, ERCP, cholecystectomy, appendectomy, colectomy or small bowel resection.
* Willing and able to give informed consent in either English or Spanish.

Exclusion Criteria:

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Patients not meeting entry criteria above.
* Refusal to give informed consent.
* Coagulopathy (INR > 2 and/or platelet count < 100,000.
* White Blood Cell count < 5,000/mm3
* Arrhythmia
* Serum creatinine > 2 mg/dl
* Prior known or suspected nasal obstruction.
* Known or suspected Zenker's diverticulum of esophagus, esophageal stricture, head/neck radiation therapy, hereditary telangiectasis, esophageal varices, cirrhosis.
* Anticoagulant usage such as heparin or Plavix

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Total time of the return of normal pharyngoesophageal function | During the last 15 minutes of general anesthesia use
  Our primary objective is to determine the timing of the return of normal pharyngoesophageal function upon withdrawal of general anesthesia.

SECONDARY OUTCOMES:
Number of participants with normal pharyngoesophageal function. | During the last 15 minutes of general anesthesia use
  Correlation of the return of normal pharyngoesophageal function with other markers generally used by Anesthesia staff to indicate a safe time for removal of endotracheal tubes.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Rogers, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No